CLINICAL TRIAL: NCT00920712
Title: Study of the Chinese Prescription Weiqi Decoction on Chronic Atrophic Gastritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHTCM-001
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2009-08

CONDITIONS: Gastritis
Keywords: chronic atrophic gastritis; Traditional Chinese Medicine
MeSH Terms: conditions — Gastritis; Gastritis, Atrophic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weiqi decoction (Experimental)
  Interventions: Drug: Weiqi decotion
- low dose of Weiqi decoction (Placebo Comparator)
  Interventions: Drug: Weiqi decotion

INTERVENTIONS:
Drug: Weiqi decotion — Decoction ,two times a day

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the Chinese prescription Weiqi decoction on Chronic Atrophic Gastritis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Atrophic Gastritis
* Male of female patients between 18-65 years old
* Written informed consent

Exclusion Criteria:

* Combine with malignant pathology on epithelial dysplasia of gastric mucosa
* Combine with duodenal ulcer or gastric ulcer
* Combined with severe heart, gallbladder, kidney, endocrine system, hemopoietic system or nervous system disease.
* Pregnancy or breast feeding women, or unwilling to have contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Symptoms and conditions of tongue and pulse,the gastroscopy and pathological change | 12 weeks

SECONDARY OUTCOMES:
Indicates of liver and renal function | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xie Jianqun, Phd, Study Director — Shanghai University of Chinese Medicine
Locations (1):
- Longhua hospital, Shanghai, Shanghai Municipality, China